CLINICAL TRIAL: NCT03365999
Title: Comparative Study of the Efficiency of Oral Tranexamic Tcid vs. Oral Tminocaproic Acid to Reduce Blood Loss and Transfusion After Total Knee Replacement. A Prospective, Randomized, Double Blinded Controlled Clinical Trial.
Brief Title: Oral Tranexamic Acid vs. Oral Aminocaproic Acid to Reduce Blood Loss and Transfusion After Total Knee Replacement.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, FELIX VILCHEZ CAVAZOS, Professor of Orthopedics and Traumatology, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OR17-00014
Record Dates: First submitted 2017-11-17; First posted 2017-12-08 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Knee Osteoarthritis; Blood Clot; Transfusion Related Complication; Blood Loss
MeSH Terms: conditions — Osteoarthritis, Knee; Thrombosis; Hemorrhage | interventions — Tranexamic Acid; Aminocaproic Acid

STUDY DESIGN:
Intervention Model Description: Two study groups will be generated, each consisting of 40 research subjects, randomly each recipient will receive 3 doses of one of the two study drugs (tranexamic acid or aminocaproic acid). The group to which the patient belongs will be assigned through a computer program, the patient will not know to which group he belongs or what medication he will receive. The patients will be extracted from the external traumatology clinic.
Who Masked: Participant
Masking Description: Prior to being included in the study, the patient will be mentioned the times when he will receive the medication as well as the dosage of administration (which is the same for each of the two medications). The patient will not know what medication is being administered to him / her. no time The pills will be given to you in a medicine cup without access to any information legend.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oral Tranexamic Acid (Active Comparator): Tranexamic acid will be administered orally three times (administering 2 tablets each time). In the case of tranexamic acid tablets are 650 mg each.
  The first administration will be two hours before the induction of anesthesia, the second 6 hours post-surgery and the third 12 hours after surgery. All by oral administration with a drink of water. The medicines will be administered with a volume of 40 ml of water.
  For the tranexamic acid a total dose of 3.9 grams (6 tablets) divided between the 3 administrations (1.3 grams each, ie 2 tablets of 650 mg) will be administered.
  Interventions: Drug: Oral Tranexamic Acid
- Oral Aminocaproic Acid (Experimental): Aminocaproic acid will be administered orally three times (administering 2 tablets each time). In the case of aminocaproic acid tablets are 500 mg each.
  The first administration will be two hours before the induction of anesthesia, the second 6 hours post-surgery and the third 12 hours after surgery. All by oral administration with a drink of water. The medicines will be administered with a volume of 40 ml of water.
  For the aminocaproic acid, a total dose of 3 grams (6 tablets) divided between the 3 administrations (1 gram each, ie 2 tablets of 500 mg) will be administered.
  Interventions: Drug: Oral Aminocaproic Acid

INTERVENTIONS:
Drug: Oral Tranexamic Acid — Patients undergoing total knee replacement who will receive three doses of tranexamic acid administered orally (1 prior to surgery and 2 subsequent to surgery).
  Arms: Oral Tranexamic Acid
Drug: Oral Aminocaproic Acid — Patients undergoing total knee replacement who will receive three doses of aminocaproic acid administered orally (1 prior to surgery and 2 subsequent to surgery).
  Other Names: Amicar
  Arms: Oral Aminocaproic Acid

SUMMARY:
This study compares two oral medications (tranexamic acid and aminocaproic acid) as hemostatic agent administered in patients undergoing total knee replacement.

DETAILED DESCRIPTION:
Background

Total knee arthroplasty is the most common orthopedic procedure in knee surgery for the treatment of degenerative diseases such as OA and rheumatoid arthritis (RA), with nearly 700,000 procedures performed in 2012 in the USA. The TKA frequently results in a significant loss of blood in a post-operative manner, which is estimated at more than 1500 ml (Hart et al., 2014). It has been reported that about 20 to 50% of patients under an TKA require a transfusion of allogenic blood. Even so, transfusion is associated with high costs, a high rate of hemolytic and non-hemolytic transfusion reactions, transmission of infectious diseases, high incidence of fluid overload and higher rates of post-operative morbidity and mortality. It has been reported in previous studies that the cost related to the transfusion of a single globular package reaches 1200 dollars (Bierbaum et al., 1999).

Tranexamic acid (AXA) and aminocaproic acid (EACA) are synthetic drugs derived from Lysine that competitively inhibit the lysine receptors in the plasminogen and plasmin activating molecules, preventing the premature dissolution of the clot. These can be administered orally, intravenously or topically. Previous studies of systematic reviews have concluded that the topical and intravenous forms of tranexamic acid significantly decrease bleeding after an TKA (Churchill et al., 2016).

Regarding the administration routes of the drugs in the intravenous form, cases of severe anaphylaxis and / or septic shock have been observed during its administration. The topical form carries the theoretical risk of increasing the rate of periprosthetic infections due to contamination of the needle and could cause sepsis. In the same way, the effects of topical application on the duration of the cement used in the prosthesis has not been determined in studies with long-term follow-up.

There are 3 forms of presentation for the administration of tranexamic acid (oral, topical and intravenous), however the ideal route for its administration remains controversial. Yuan et al. (2017) conducted a study comparing the 3 routes of administration of tranexamic acid during the total replacement of the unilateral primary knee, finding that the three routes are effective in reducing blood loss and the rate of transfusion. In the same way, the oral route of administration proved to be equivalent or even more effective in the total replacement of the knee and hip to reduce blood loss. Similarly from a cost-benefit point of view it has also proven to be superior.

Stabilizing the clot, antifibrinolytic drugs reduce perioperative blood loss and the need for transfusions. The use of AXA has recently become a popular strategy implemented by orthopedic surgeons in order to reduce blood loss and the rate of transfusions (Kim et al., 2014). An increase in postoperative bleeding has been described after the removal of the pneumatic tourniquet in the total knee replacement (TKR), which is attributed to the activation of the fibrinolytic system in the first hours after surgery (Jansen et al., 1999). This effect is positive by reducing the risk of a thromboembolic event associated with an orthopedic procedure, however it increases the risk of post-operative bleeding which increases the chances of requiring a transfusion (Spahn and Cassut, 2000).

Medications that reduce hyperfibrinolysis can be administered to reduce blood loss (Spahn and Cassut, 2000). ATX and AAC are two drugs that can be used to prevent perioperative blood loss in TKR and other orthopedic procedures (Yamasaki et al., 2005, Bennett-Guerrero et al., 1997).

The oral administration of antifibrinolytic drugs decreases the risk of developing anaphylaxis that occurs more frequently with the use of the intravenous route. For AXA it has been shown that both intravenous and oral routes are effective in reducing blood loss and the rate of transfusion.

AAC is an effective antifibrinolytic when administered and is less expensive than the AXA so its use by oral route would reduce the risk of anaphylactic reactions in addition to reducing the cost of treatment. It has an average cost in its use of 2.70 dollars per surgical procedure in its intravenous form, compared to 40 dollars per surgery with the use of tranexamic acid in total hip replacement.

At the moment there are no comparative studies of the efficacy of tranexamic acid and aminocaproic acid administered orally for the reduction of bleeding and transfusion index in patients undergoing total knee replacement.

HYPOTHESIS

There are no significant differences in blood loss, transfusion index and hemoglobin levels in patients undergoing total knee prostheses treated with tranexamic acid or aminocaproic acid orally.

OBJETIVES

General objective

1. To compare the effect of oral aminocaproic acid as a hemostatic agent against oral tranexamic acid administered preoperatively and postoperatively in patients undergoing elective surgery of total knee replacement due to primary osteoarthrosis.

Specific objectives

1. Selection and randomization of patients.
2. Performing total knee replacement surgery and administration of AAC or AXA according to randomization and the methodology established in this protocol
3. Establishment of a protocol for the administration of aminocaproic acid orally for its use as a hemostatic agent in elective surgery of total knee replacement.
4. Determination of blood loss, transfusion index, decrease in hemoglobin and hematocrit levels, drainage volume, intrahospital stay, analogous visual scale, SF-12 scale, thromboembolic complications and complications related to the wound between tranexamic acid and the aminocaproic acid, both orally, in each group in the pre, peri and post-operatively established times and compare them statistically.
5. Determine and record the possible complications and side effects observed with the use of both drugs included in the study.
6. Determine the cost and monetary savings associated with the administration of each drug.
7. Comparison and statistical analysis of the results between the study groups.

5.- METHODOLOGY

Type of study: Controlled clinical trial.

Study design: Experimental, longitudinal, comparative, prospective and blind.

Approximate duration of the study: 18 months

Type of population and sample size: A total of 80 patients undergoing elective surgery of total knee replacement due to unilateral primary gonarthrosis (40 patients per group) will be included.

Investigation Site: Patients will be recruited from Consultation No. 15 of the Orthopedics and Traumatology Service of the University Hospital "Dr. José Eleuterio González "of the U.A.N.L. and the surgery will be carried out in the Surgical Therapeutics Department of the 5th floor of the University Hospital of the U.A.N.L.

Randomization mode: 80 sealed envelopes in which the group to which the patient belongs will be prepared prior to the start of the study. The patient will not know the group he will belong to until the moment of revealing the final results of the study.

Recruitment Methodology: Each patient who is admitted for elective surgery of total knee replacement will be invited to participate voluntarily in the study. The principal investigator or one of the co-investigators will be responsible for thoroughly explaining the details of the study, including the potential benefits and risks thereof, as well as answering any doubts that may arise, if the patient agrees to participate they will be asked to sign the informed consent in the presence of two witnesses and a note will be made in the clinical file where their inclusion in the study will be registered, in the same way a copy of the consent will be given to the patient. For the purposes of the study, it will not be necessary to identify the patient, only their gender and age.

The Head of the Anaesthesiology Service will be informed about the implementation of the protocol for the training in the management of the drugs to be administered in this protocol, to the nursing staff and residents of anesthesiology. The study population will be divided into 2 groups: 1. Tranexamic Acid Group and 2. Aminocaproic Acid Group with a total of 80 patients (40 patients per group). The randomization process will be randomized by means of a statistical software.

The surgeries of all the groups will be performed with the same surgical technique, using a total knee prosthesis model Vanguard, brand Biomet (Warsaw, IN), stabilized earlier. The patients will be operated by 3 subspecialists in joint knee surgery, professors of the Orthopedics and Traumatology Service of the University Hospital "Dr. José Eleuterio González "as the main surgeon and as surgical assistants, the resident physicians of Orthopedics and Traumatology who are rotating through the knee module or joint replacement.

Surgical technique

Previous epidural neuraxial block, prophylactic dose of antibiotic (Vancomycin 1 gr IV dissolved in 250 ml of 0.09% NaCl Physiological Solution to pass in two hours, administered 150 minutes prior to the surgical procedure), using tourniquet at 100mmHg over the systolic pressure of the patient and previous protocol of asepsis and antisepsis (washing with 2% chlorhexidine the entire limb for 6 minutes and with duraprep® the area of the knee immediately prior to the initial incision) and placement of sterile fields. An insall type, medial parapatellar surgical approach will be performed and the conventional surgical technique will be followed for the placement of a two-compartment knee prosthesis.

Subsequently, the wound will be closed by layers (capsule, subcutaneous cellular tissue and skin) in both groups. A 1/8 drenovack will be placed, fixed to the skin, which will be pinched for 1 hour and removed 48 hours after surgery. Thromboprophylaxis will be initiated with low molecular weight heparin 6 hours after the end of surgery. In the postoperative period, all patients with Hb levels of less than 8 mg / dl or with anemic syndrome clinical data will be transfused.

Drug administration protocol:

The sealed envelope will be opened on the preoperative day to identify which experimental group the patient belongs to and the oral administration of the medication will be included within the preoperative indications of the patient.

Each patient will receive 3 doses of the drug to be evaluated according to the group to which it corresponds (1 preoperative dose and 2 postoperative doses). The protocol for the pre and post-operative administration of the drugs will be as follows:

Medications: tranexamic acid (Lysteda, Pierre Fabre Mexico) or aminocaproic acid (Amikar, Wyeth), as appropriate, will be administered orally three times (administering 2 tablets each time). In the case of aminocaproinco tablets are 500 mg each and in the case of tranexamic acid are 650 mg each.

The first administration will be two hours before the induction of anesthesia, the second 6 hours post-surgery and the third 12 hours after surgery. All by oral administration with a drink of water. The medicines will be administered with a volume of 40 ml of water.

For the aminocaproic acid, a total dose of 3 grams (6 tablets) divided between the 3 administrations (1 gram each, ie 2 tablets of 500 mg) will be administered. For aminocaproic acid a total dose of 3.9 grams (6 tablets) divided between the 3 administrations (1.3 grams each, ie 2 tablets of 650 mg) will be administered.

Parameters to be evaluated

The general data of the patient will be obtained: age, gender, weight, height, body mass index and personal history, time of evolution of knee osteoarthritis and previous treatments, classification of osteoarthritis in the Kellgreen and Lawrence scale, femoro-tibial angle (APPENDIX 1). Pre-operative hemoglobin and hematocrit levels will be measured. As well as, at 6 a.m. (24, 48 and 72 hours postsurgery). The expense for the drenovack will be measured / quantified at 6am (24 and 48 hours postsurgery). The transfusion rate will be measured, according to the level of hemoglobin described before. Finally the functional scales; Analogous visual scale (EVA); at 24, 48 and 72 hours and the SF-12 scale (ANNEX 2) (Vilalgut et al., 2005; Alonso et al., 1998; Ware et al., 1996; Gandek et al., 1998) in the preoperative day and in the 3rd postoperative day (hospital discharge).

They will also obtain and analyze the amount of bleeding during surgery, the surgical time and peri and post-operative complications.

Intrahospital follow-up

Anticoagulation will be initiated with Heparin 5000 U.I subcutaneously 6 hours after the surgical procedure, and once in the hospitalization area the quantification of the drenovack expense will begin, a blood biometry and the administration of intravenous analgesia will be requested. On the day after the surgical procedure, the first surgical wound healing will be performed and the patient will start walking assisted by the doctor (this represents the normal post-operative management protocol of the patient undergoing a total knee replacement in our service).

Patient's discharge

It will be discharged by medical indication to the patient on the third post-operative day, if there is no type of contraindication, with indications of discharge in medical prescription and follow-up by the external consultation after two weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years
2. Total replacement of the primary knee due to primary Osteoarthrosis
3. Two-compartment prosthesis
4. Unilateral procedure
5. Cemented prosthesis
6. Desire to participate voluntarily in the study and signature of informed consent
7. Pre-operative assessment with result between ASA I, ASA II or ASA III performed and annexed in the clinical file either by the Department of Internal Medicine, Cardiology or Anesthesiology of our hospital.
8. Possibility for oral administration of the drug.

Exclusion Criteria:

1. History of thrombotic or embolic event in the last 6 months
2. Clinical history of coagulopathy
3. Previous surgeries in the knee to intervene
4. Patients who have received aspirin, platelet or cumarinic antiplatelet agents in the week prior to surgery or NSAIDs two days prior to surgery.
5. History of myocardial infarction, arteriopathy or unstable angina in the 12 months prior to surgery.
6. Those patients whose preoperative assessment corresponds to an ASA IV or the procedure is contraindicated in its preoperative assessment.
7. Total revision knee replacement
8. Total replacement of tumoral knee
9. Total bilateral knee replacement
10. Cognitive deficit
11. Patients who meet the inclusion criteria but do not wish to participate in the study
12. Patients with a diagnosis of Terminal Chronic Kidney Disease or with a serum creatinine higher than 1.47 mg / dl in the preoperative laboratories.
13. Patients with inability to ingest the drug orally.
14. Patients who are pregnant or breast-feeding or who are taking oral contraceptives.
15. Seizure history
16. Hypersensitivity to the active substance or to any of the excipients.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Total blood loss (TBL) | The third day postoperative,at the time of obtaining the result of the hematocrit of 72 hours.
  Total blood loss 72 hours after surgery,The Gross and Nadler formula was used to calculate TBL. TBL = patient's blood volume (PBV) x (Hctpre - Hctpost)/Hctave (Hctpre = the initial pre-operative Hct level, Hctpost = the Hct on the morning of POD3). PBV = k1 x height (m) + k2 x weight (kg) + k3 (k1 = 0.3669, k2 = 0.03219, and k3 = 0.6041 for men; and k1 = 0.3561, k2 = 0.03308, and k3 = 0.1833 for women, Hctave = the average of the Hctpre and Hctpost)
External blood loss (EBL) | On the second postoperative day (48 hours), when removing the surgical drainage.
  External blood loss (EBL) was estimated by adding the intraoperative bleeding and the blood in the drain collectors upon removal after 48 hours
Hidden blood loss (HBL) | The third day postoperative
  was defined as Total blood loss minus External blood loss

SECONDARY OUTCOMES:
Chage in Hematocrit level | Hematocrit levels will be measured at 24, 48 and 72 hours postsurgery
  Hematocrit levels obtained in 3 samples taken at different times postsurgery
Drainage quantification | Drainage quantification will be registered at 24 and 48 hours postsurgery
  Drainage will be quantified in ml at 2 different times postsurgery
Therapeutic effect on visual analog scale | The third day postoperative
  The pain Visual Analog Scale is a unidimensional measure of pain intensity. The scale is most commonly anchored by "no pain " (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (scale of 10). It will be assessed as a numeric scale from 0 to 10.
Change in Hemoglobin level | Hemoglobin levels will be measured at 24, 48 and 72 hours postsurgery
  Hemoglobin levels obtained in 3 samples taken at different times postsurgery
Complications | at 24, 48 and 72 hours, 7 days, 4 and 6 weeks.
  Complications related to the surgery or to the administration of the study medication
Transfusion rate | at 24, 48 and 72 hours, 7 days, 4 and 6 weeks.
  Need to administer globular packages following the indications of transfusion haemaglobin (Hb) of 8 g/dl in patients free of cardiovascular disease and Hb of 9 g/dl in patients with established cardiovascular disease or cardiovascular risk factors with symptoms of anaemia (defined as bad mental status, palpitation, or shortness of breath not due to othercauses). Hb below 10 g/dl in patients with poor clinical tolerance of lower values was also an indication for transfusion. Symptoms of poor clinical tolerance of lower values were signs of hypoxia such as tachycardia, dyspnoea or syncope or drainage of more than 1 l of blood in the first 24 hours.
Intraoperative blood loss | Immediately after the end of the surgery
  Intra-operative blood loss was calculated using the difference between the weights of the used gauze and the original unused gauze (25 cm x 25 cm, monolayer, weight of 30 grams), in addition to the blood volume accumulated in suction bottles subtracting the volume of saline solution during the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Felix Vilchez-Cavazos, MD PhD, Principal Investigator — UANL
Locations (1):
- Facultad de Medicina UANL, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No
Sharing information has not been discussed with the ethics committee, it is necessary to define the need to share information relative to patients in order to perform and establish specific actions.

REFERENCES:
- [Result] Boese CK, Centeno L, Walters RW. Blood Conservation Using Tranexamic Acid Is Not Superior to Epsilon-Aminocaproic Acid After Total Knee Arthroplasty. J Bone Joint Surg Am. 2017 Oct 4;99(19):1621-1628. doi: 10.2106/JBJS.16.00738. PMID 28976426
- [Result] Harper RA, Sucher MG, Giordani M, Nedopil AJ. Topically Applied Epsilon-Aminocaproic Acid Reduces Blood Loss and Length of Hospital Stay After Total Knee Arthroplasty. Orthopedics. 2017 Nov 1;40(6):e1044-e1049. doi: 10.3928/01477447-20170925-07. Epub 2017 Oct 3. PMID 28968480
- [Result] Hobbs JC, Welsby IJ, Green CL, Dhakal IB, Wellman SS. Epsilon Aminocaproic Acid to Reduce Blood Loss and Transfusion After Total Hip and Total Knee Arthroplasty. J Arthroplasty. 2018 Jan;33(1):55-60. doi: 10.1016/j.arth.2017.08.020. Epub 2017 Aug 24. PMID 28939033
- [Result] Churchill JL, Puca KE, Meyer E, Carleton M, Anderson MJ. Comparing epsilon-Aminocaproic Acid and Tranexamic Acid in Reducing Postoperative Transfusions in Total Knee Arthroplasty. J Knee Surg. 2017 Jun;30(5):460-466. doi: 10.1055/s-0036-1593362. Epub 2016 Oct 3. PMID 27699724
- [Result] Banerjee S, Issa K, Pivec R, McElroy MJ, Khanuja HS, Harwin SF, Mont MA. Intraoperative pharmacotherapeutic blood management strategies in total knee arthroplasty. J Knee Surg. 2013 Dec;26(6):379-85. doi: 10.1055/s-0033-1353992. Epub 2013 Aug 16. PMID 23955184
- [Result] Sepah YJ, Umer M, Ahmad T, Nasim F, Chaudhry MU, Umar M. Use of tranexamic acid is a cost effective method in preventing blood loss during and after total knee replacement. J Orthop Surg Res. 2011 May 21;6:22. doi: 10.1186/1749-799X-6-22. PMID 21600028
- [Result] Camarasa MA, Olle G, Serra-Prat M, Martin A, Sanchez M, Ricos P, Perez A, Opisso L. Efficacy of aminocaproic, tranexamic acids in the control of bleeding during total knee replacement: a randomized clinical trial. Br J Anaesth. 2006 May;96(5):576-82. doi: 10.1093/bja/ael057. Epub 2006 Mar 10. PMID 16531440
- [Result] Ahlberg A. Diffusion of epsilon aminocaproic acid to the joints. Proc Soc Exp Biol Med. 1970 Sep;134(4):988-9. doi: 10.3181/00379727-134-34927. No abstract available. PMID 4195730